CLINICAL TRIAL: NCT07033741
Title: Predictors and Process Moderators of EMDR Therapy for Depressive Symptoms: Protocol for a Real-world Prospective Observational Study
Brief Title: Predictors and Process Moderators of EMDR Therapy for Depressive Symptoms
Acronym: PROCESS-EMDR
Status: Recruiting | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, luca ostacoli, Full Professor, University of Turin, Italy
Other Study IDs: PROCESS-EMDR/0565145
Record Dates: First submitted 2025-04-30; First posted 2025-06-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Depression, Anxiety; Post-traumatic Stress Symptoms; Dissociation; Psychotherapy Research and Outcome Measures
Keywords: Eye Movement Desensitization and Reprocessing; depressive symptoms; predictors; moderators; psychotherapy; study protocol
MeSH Terms: conditions — Depression; Anxiety Disorders; Dissociative Disorders | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EMDR Therapy Group: Participants receive Eye Movement Desensitization and Reprocessing (EMDR) therapy in accordance with standardized clinical protocol. The assessment of clinically significant symptoms will be conducted using validated screening tools and diagnostic measures aligned with the study 's objectives. The initial session (Timepoint 0a [T0a]) will consist of a thorough baseline evaluation, in which participants will fill out a set of baseline self-report questionnaires. A second baseline assessment (T0b) will take place after the completion of four therapy sessions, focusing on changes in emotional regulation, personal beliefs, attachment style, and the processing of traumatic memories. Both the patient and therapist will evaluate the therapeutic alliance at T0b, offering insights into the evolving dynamics of the therapeutic process. After baseline assessments (T0a and T0b), additional assessments will occur at six (T6), twelve (T12), with a maximum follow-up period of eighteen months (T18).
  Interventions: Behavioral: EMDR

INTERVENTIONS:
Behavioral: EMDR — The EMDR process follows an eight-phase protocol that includes (1) history taking: gathering patient's background information and planning treatment, (2) preparation: preparing the patient for processing target, (3) assessment: accessing target of the traumatic memories, (4) desensitization: processing target memories using dual task , (5) installation: strengthening the alternative positive cognition, (6) body scan: noting any physical sensations related to the target memory, (7) closure: ensuring patient's stability at the end of the session, and (8) revaluation: assessing effectiveness of the session and future planning.

SUMMARY:
The goal of this clinical trial is to evaluate which factors influence the effectiveness of Eye Movement Desensitization and Reprocessing (EMDR) therapy for depressive symptoms in real-world settings in Italy.

The main questions the study seeks to answer are:

* Which key factors influence EMDR outcomes in terms of mediators, moderators, and predictors of its effectiveness for depressive symptoms?
* Do lower levels of individual psychological functioning at baseline, including high co-occurrence of personality domains and pathogenic personal beliefs, predict the effects of EMDR in treating depressive symptoms?
* Are baseline psychological comorbidities (anxiety, dissociation, post-traumatic symptoms, emotional dysregulation, and sleep difficulties) and the quality of the therapeutic alliance related to the effectiveness of EMDR therapy for depressive symptoms? Participants will be both therapists and patients.
* Eligible therapists must be certified members of the EMDR Italian National Association to ensure adherence to established standards in the practice of EMDR therapy and consistency in therapeutic delivery. Therapists will identify patients from their routine clinical practice who meet the study inclusion criteria and facilitate their enrollment.
* Eligible patients must meet the following criteria:

  1. Being 18 years of age or older.
  2. being able to give informed consent.
  3. presenting clinically significant symptoms in at least one of the following domains: anxiety, depression, dissociative, or post-traumatic stress symptoms.

Individuals presenting with severe neurological impairment or other severe psychiatric conditions were excluded.

Researchers will combine data from multiple N-of-1 trials (N-of-1 or single-subject clinical trials studies) using a Bayesian multilevel random-effects meta-analysis and meta-regression to generate robust estimates of treatment efficacy.

ELIGIBILITY:
Participants:

Therapist

* Inclusion Criteria:
* certified members of the Italian Eye Movement Desensitization and Reprocessing (EMDR) Association
* Exclusion Criteria:
* inability or unwillingness to comply with study protocols or schedules Patient
* Inclusion Criteria:
* age 18 years or older
* capacity of providing informed consent
* presenting with clinically significant symptoms in at least one of the following domains: anxiety, depression, post-traumatic stress symptoms, or dissociative symptoms.
* Exclusion Criteria:
* history of psychotic symptoms or schizophrenia
* dementia
* severe personality disorders
* a serious, unstable medical condition
* acute suicidality that needs hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include members of the Italian National EMDR Association who are in private practice. Each therapist will select one of their patients to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Monitoring depressive symptoms | Baseline, during the intervention, 6 months, 12 months, through study completion (an average of 18 months)
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report tool used to measure depressive symptoms. Participants rate the frequency of symptoms over the previous 2-week period on a scale from 0 ("not at all") to 3 ("nearly every day"), with total scores indicating no symptoms (0-5 points), mild symptoms (6-10 points), moderate symptoms (11-15 points), or severe symptoms (greater than 15 points).
Depressive symptoms | Baseline, 6 months, 12 months, at study completion (an average of 18 month)
  The Beck Depression Inventory (BDI-II) is a 21-item self-report instrument that assesses the severity of depressive symptoms based on DSM-IV criteria. The total score ranges from 0 to 63, with higher scores indicating greater levels of depression. A score above 13 is considered the cut-off for depressive symptoms (14-19: mild depression; 20-28: moderate depression; ≥29: severe depression).

SECONDARY OUTCOMES:
Personal beliefs | Baseline, at study completion (an average of 18 month)
  The Personal Beliefs Scale-Revised (PBS-R) is a 44-item self-report measure designed to evaluate maladaptive personal beliefs across domains such as self-worth, interpersonal relationships, and personal agency. Respondents first indicate whether each belief applies to them by selecting "yes" or "no". For beliefs marked as applicable, participants then rate the degree to which each belief is problematic or distressing on a 4-point Likert scale, ranging from 1 ("not at all") to 4 ("very problematic").
Personality domains | Baseline, at study completion (an average of 18 month)
  The Personality Inventory for DSM-5 - Brief Form (PID-5-BF) is a 25-item self-report measure designed to assess five personality trait domains: negative affect, detachment, antagonism, disinhibition, and psychoticism. Each domain consists of 5 items rated on a 4-point scale ranging from 0 ("very false or often false") to 3 ("very true or often true"). The total score ranges from 0 to 75, with higher scores indicating greater personality dysfunction, while individual domain scores range from 0 to 15. Consistently high scores in a particular domain may indicate significant and challenging areas for the patient that may warrant further assessment, treatment, or follow-up.
Anxiety symptoms | Baseline, during the intervention, 6 months, 12 months, at study completion (an average of 18 month)
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report instrument designed to measure the frequency of generalized anxiety symptoms over the previous 2-week period on a scale from 0 ("not at all") to 3 ("nearly every day"). Total scores indicate no symptoms (0-5 points), mild symptoms (6-10 points), moderate symptoms (11-15 points), or severe symptoms (greater than 15 points).
Dissociative symptoms | Baseline, 6 months, 12 months, at study completion (an average of 18 months)
  The Dissociative Experiences Scale (DES-II) is a 28-item, self-report assessment tool designed to measure dissociative experiences, including emotional involvement, depersonalization, derealization, compartmentalization, and amnesia. Each item on the scale evaluates the proportion of time an individual experiences the specific symptom. The overall score is calculated as the average of all item scores, ranging from 0% ("never") to 100% ("always").
Assessing dissociative phenomena | At second baseline timepoint (after four therapy sessions), after six months from the first baseline assessment, after twelve months from the first baseline assessment, and at end of data collection (after eighteen month)
  The Multidimensional Dissociation Inventory (MDI) is a 30-item self-report tool designed to assess dissociative phenomena across six domains: Disengagement, Depersonalization/Derealization, Emotional Constriction, Memory Disturbance, and Identity Dissociation. Each item is rated on a 5-point Likert scale ranging from 0 ("never") to 4 ("very often").
Therapeutic progress and outcomes for individuals | Baseline, 6 months, 12 months, through study completion (an average of 18 months)
  The Progress in Treatment Questionnaire - Patient (PITQ-p) is a 32-item self-report measure completed by patients, focusing on their ability to manage emotions, symptoms, relationships, safety, and overall well-being. Patients report the percentage of time they exhibit specific behaviors during the previous week, using a scale ranging from 0% ("never") to 100% ("always"). Item.
  The Progress in Treatment Questionnaire - Therapist (PITQ-t) is a 29-item measure designed to assess the percentage of time patients demonstrate treatment target behaviors over the prior 6 months. Each item is rated on a scale ranging from 0% ("never") to 100% ("always"). The questionnaire includes six specific items (items 24-29) for patients exhibiting dissociative self-states. Higher scores reflect greater adaptive functioning. The PITQ-t helps therapists evaluate multiple areas of patient functioning, providing a structured approach to monitoring progress and refining treatment plans.
Post-traumatic Stress symptoms | Baseline, 6 months, 12 months, at study completion (an average of 18 month)
  The Post-traumatic Stress Disorder Checklist (PCL-5) is a 20-item self-report assessment designed to evaluate the presence and severity of PTSD symptoms. Each item is rated on a 5-point Likert scale, where 0 indicates the absence of symptoms and 4 indicates extreme severity. The items of the PCL-5 are designed to be aligned with the DSM-5 diagnostic criteria for PTSD. The total score ranges from 0 to 80, with higher scores indicating greater levels of PTSD symptoms. A cutoff score of 33 is considered a reasonable threshold for provisional PTSD diagnosis.
Emotion regulation | Baseline, 6 months, 12 months, at study completion (an average of 18 months)
  The Difficulties in Emotion Regulation Scale (DERS) is a 36-item, self-report questionnaire to assess how individuals perceive and manage relevant difficulties in their emotional experiences. It is related to various aspects of emotion regulation, including acceptance of emotional responses, impulse control, emotional clarity, and the use of emotion regulation strategies. Respondents are asked to rate their agreement on a 5-point Likert scale ranging from 1 ("strongly disagree") to 5 ("strongly agree").
Quality of sleep | Baseline, 6 months, 12 months, at study completion (an average of 18 month)
  The Mini Sleep Questionnaire (MSQ) is a 10-item self-report instrument designed to assess sleep quality and sleep disorders. Each item is rated on a 7-point Likert scale, ranging from 1 ("never") to 7 ("always"). Four levels of sleep quality are identified: 10-24 (good sleep quality), 25-27 (mild sleep difficulties), 28-30 (moderate sleep difficulties), and ≥31 (severe sleep difficulties).
Therapeutic alliance | Baseline, 6 months, 12 months, at study completion (an average of 18 months)
  The Working Alliance Inventory (WAI) is a 36-item self-report measure designed to assess the quality of the therapeutic alliance available in both therapist (WAI-T) and patient (WAI-P) versions. The scale evaluates three fundamental dimensions of the therapeutic relationship: goals (agreement on therapy objectives), tasks (agreement on the steps or methods to achieve these goals), and bond (the emotional connection and mutual trust between therapist and patient). Each item is rated on a 7-point Likert scale ranging from 1 ("never") to 7 ("always"), with higher scores reflecting a stronger working alliance. Subscale scores provide detailed insights into the specific components of the alliance, while the total score represents the overall strength of the therapeutic relationship.
  The study also includes study-specific evaluation forms designed to gather targeted information on therapeutic processes and clinical outcomes.

OTHER OUTCOMES:
Exposure to traumatic or stressful life events | Baseline
  The Life Stressor Checklist-Revised (LSC-R, Wolfe et al., 2012), is a self-report measure used to assess exposure to traumatic or stressful life events throughout the lifespan, such as natural disasters, interpersonal violence, and the sudden death of a loved one. Respondents use a dichotomous response format (yes/no) to indicate whether they have experienced each event. For endorsed events, participants provide additional details, including the age of occurrence, whether they felt in harm's way or helpless ("yes" or "no"), and rate the event's impact and associated emotional distress on a 5-point Likert scale (1 = "not at all" to 5 = "extremely"). Respondents are also asked to identify up to three events that currently have the greatest impact on their lives. The LSC-R is widely used in clinical and research contexts to evaluate the cumulative effects of life stressors and their psychological impact.
Compassion | Baseline, during the intervention, 6 months, 12 months, at study completion (an average of 18 months)
  The Compassionate Action and Engagement Scales (CAES) is a self-report instrument designed to assess three key dimensions of compassion: (1) the compassion one experiences for others, (2) the compassion one perceives from others, and (3) self-compassion. The scales are based on a standard definition of compassion as "a sensitivity to suffering in self and others, coupled with a commitment to alleviate and prevent it". The instructions for each scale define compassion and invite participants to reflect on their responses when confronted with their own suffering, the suffering of others, or the experience of compassion from others. Responses are recorded using a 10-point Likert scale ranging from "never" to "always". Higher scores reflect greater levels of sensitivity and commitment within each dimension of compassion.
Experience of Mindfulness | Baseline, 6 months, 12 months, at study completion (an average of 18 months)
  The Philadelphia Mindfulness Scale (PHLMS-I) is a 20-item self-report inventory designed to measure two core components of mindfulness: awareness (attentiveness to present-moment experiences) and acceptance (a non-judgmental attitude toward thoughts and emotions). Each subscale comprises 10 items rated on a 5-point Likert scale ranging from 1 ("never") to 5 ("very often"), reflecting the frequency of the subjective experiences. Subscale scores are calculated as the sum of their respective items, with higher scores indicating greater mindfulness abilities.
Evaluating adult attachment style | Baseline, at study completion (an average of 18 months)
  The Relationships Questionnaire (RQ), is a 4-item self-report tool used to assess an individual's adult attachment style. Respondents rate their agreement or disagreement with four statements on a 7-point Likert scale ranging from 1 ("strongly disagree") to 7 ("strongly agree"). The RQ identifies whether an individual has a secure, anxious, or avoidant attachment style and provides insights into how they approach and experience interpersonal relationships.
Evaluating difficulties during memory processing with EMDR sessions | During the intervention, 6 months, 12 months, through study completion (an average of 18 months)
  The Processing Difficulties Scale (PDS) is a 17-item self-report instrument designed to evaluate challenges encountered during memory processing in EMDR therapy, following the standard protocol. Clinicians rate each item on a 5-point Likert scale ranging from 0 ("never") to 4 ("always"), assessing specific processing styles. These styles include indicators of poor processing characterized by a lack of generalization, effective general processing, unproductive emotional processing, and signs of loss of dual attention during sessions. The PDS provides valuable insights into the quality and style of processing, aiding clinicians in identifying potential barriers to therapeutic progress.
Changing in memory processing | During the intervention, 6 months, 12 months, at study completion (an average of 18 months)
  The Recalled Memory Evaluation is a 14-item self-report instrument designed to assess the emotional, cognitive, and sensory aspects of memory recall after EMDR sessions (e.g., clarity, vividness, sounds, and smells). Patients rate their experience on an 11-point Likert scale ranging from 0 ("not at all") to 10 ("completely"). The form provides key insights into changes in memory processing over time, helping to share and deepen understanding of patients lived experiences of EMDR.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin, Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cotardo F, Koumantakis E, Rossini PG, Malandrone F, Berchialla P, Ostacoli L, Carletto S. Predictors and process moderators of EMDR therapy for depressive symptoms: protocol for a series of observational N-of-1 trials. Front Psychol. 2026 Jan 6;16:1688526. doi: 10.3389/fpsyg.2025.1688526. eCollection 2025. PMID 41567443